CLINICAL TRIAL: NCT05823350
Title: The Effect of Abdominal Massage on Pain and Distention in Patients Underwent Colonoscopy - A Randomized Controlled Study
Brief Title: The Effect of Abdominal Massage on Pain and Distention After Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sacide Yildizeli Topcu, Assistant Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TUTF-BAEK 2019/293
Record Dates: First submitted 2023-03-27; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Colonoscopy; Pain, Abdominal; Massage; Distension; Bowel; Patients Care; Nursing
Keywords: Abdominal massage; Colonoscopy; Abdominal pain; Patients care; Abdominal distension
MeSH Terms: conditions — Abdominal Pain; Dilatation, Pathologic

STUDY DESIGN:
Intervention Model Description: Experimental - Randomised Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The relatives of the patients were shown the video before the colonoscopy. The video consisted of visual and verbal content about colonoscopy, and the benefits and application steps of abdominal massage in pain management after the procedure.
  After the procedure, the relatives of the patients in the experimental group were asked to apply abdominal massage to their patients. During the massage application, when necessary, guidance was given to the patient's relatives about the application of the massage. In this supine position, patient's abdomen was massaged with circular movements and different techniques in the direction of the colon.
  Interventions: Other: Abdominal massage
- Control Group (No Intervention): After the procedure, the patients who were taken to their beds were asked to evaluate their pain and distension levels after the colonoscopy. The vital signs of the patients who received standard care were monitored after the procedure and were followed up for possible complications.

INTERVENTIONS:
Other: Abdominal massage — Abdominal massage after colonoscopy
  Arms: Experimental group

SUMMARY:
Aim: This study aimed to evaluate the effect of abdominal massage on pain and distention in patients who underwent colonoscopy.

Methods: This randomized controlled study was conducted between October 2019 and December 2021 with the participation of 60 patients who underwent colonoscopy in the endoscopy unit of a university hospital. Thirty patients performing abdominal massage after colonoscopy were included in the experimental group.

DETAILED DESCRIPTION:
Aim: This study aimed to evaluate the effect of abdominal massage on pain and distention in patients who underwent colonoscopy.

Methods:

Settings and Design This randomized controlled experimental study was conducted between September 2019 and September 2022 with the participation of 60 patients who underwent colonoscopy in the endoscopy unit of a university hospital.

The patients who underwent elective total colonoscopy, were accompanied by an attendant before and after the procedure, had an ASA score of ≤ 2, had no problem that would prevent the application of abdominal massage (past abdominal surgery, irritable bowel disease, diagnosis of bowel cancer, gastrointestinal or urinary ostomy, etc.), and accepted the application of abdominal massage after the procedure, were included in the study.

Patients who did not speak Turkish or didn't have any attendant who could speak Turkish, who did not want to receive abdominal massage, who couldn't learn abdominal massage or did not want to do it, and the patients for whom the procedure was not fully implemented due to reasons such as insufficient bowel preparation, were excluded from the study.

During the study's follow-up period, no complications related to colonoscopy were observed in the participating patients.

Data Collection Tools Patient information form and patient follow-up form were used for collecting research data. The patient information form included 3 questions investigating the sociodemographic characteristics of the patients (age, gender, experience of colonoscopy). The patient follow-up form contains four questions including the patients' pain and distension level after colonoscopy and abdominal massage. The level of pain and distension was evaluated with a 0-10 numerical comparison scale (Dreyer ve ark. 2015).

Data Collection The number of patients in each group was determined to be equal (30:30) by randomization carried out through the computer program called Research Randomiser. The group that received abdominal massage was accepted as the experimental group. On the day of the procedure, all patients who came to the endoscopy unit for a total colonoscopy were informed by the researcher about the study and then written and verbal informed consents were obtained from the patients.

In the control group, after the procedure, one relative was allowed to accompany each patient who was taken to the care room after the endoscopy. The patients who were taken to their beds were asked to evaluate their pain and distension levels after the colonoscopy (first evaluation). The initial pain and distension levels after the procedure were recorded on the form by the researcher. The vital signs of the patients who received standard care were monitored after the procedure and were followed up for possible complications. The pain and distension levels of the patients were evaluated again 20 minutes after the first assessment (second evaluation). After the procedure, patients who met the discharge criteria were given discharge training and they were allowed to leave the endoscopy unit after the vascular access catheter was removed.

In the experimental group, the relatives of the patients were shown the video in the preparation room before the colonoscopy. The video consisted of visual and verbal content about the definition, purposes, application, and importance of the colonoscopy, the purpose of insufflation, pain management during and after the procedure, and the benefits and application steps of abdominal massage in pain management after the procedure. The video lasted 3 minutes and 19 seconds.

After the procedure, a relative was allowed to accompany each of the experimental group patients who were taken to the care room after the endoscopy. The patients who were taken to their beds were asked to evaluate their pain and distension levels after the colonoscopy (first evaluation). The initial pain and distension levels after the procedure were recorded on the form by the researcher. Afterwards, the relatives of the patients in the experimental group were asked to apply abdominal massage to their patients. During the massage application, the patient and their relatives were observed by the researcher, and when necessary, guidance was given to the patient's relatives about the application of the massage. Liquid vaseline was used to ensure the slipperiness of the hands during the massage. In this supine position, patient's abdomen was massaged with circular movements and different techniques (kneading, vibration, efflorescence, superficial or deep strokes) in the direction of the colon.

As suggested in the literature, an abdominal massage lasted 15 minutes (Yıldırım et al. 2019). When necessary, verbal and visual guidance was provided by the researcher to ensure that the massage was performed with the correct steps and for the required time.After 5 minutes after the massage application, the researcher evaluated the patients' pain and distension levels and recorded the data on the form (second evaluation; 20 minutes after the first evaluation). After the procedure, patients who met the discharge criteria were given discharge training and they were allowed to leave the endoscopy unit after the vascular catheter was removed.

Statistical Analysis Data obtained from sixty-five patients were analyzed using the IBM SPSS 22.0 (IBM, Armonk, New York, USA) package program. Normal distribution was determined by the Kolmogorov-Smirnov test. The Mann-Whitney U test was used to compare the pain and distention scores between the two groups. Wilcoxon Signed rank test was used to compare the means of pain and distention scores within the group. The statistical significance level was accepted as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an elective total colonoscopy
* Having an attendant before and after the procedure
* ASA score ≤ 2
* Accepting the application of abdominal massage

Exclusion Criteria:

* Not knowing Turkish himself/herself or his/her attendant
* Having a problem that prevents the application of abdominal massage (past abdominal surgery, irritable bowel disease, bowel cancer diagnosis, gastrointestinal or urinary ostomy, etc.)
* Not wanting to have an abdominal massage
* Failure of the attendant to learn abdominal massage
* Inability to perform colonoscopy completely due to insufficient bowel preparation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Pain after colonoscopy | Change from abdominal pain after the colonoscopy at 20 minutes after.
  Assesment of abdominal pain after colonoscopy by using numerical pain scale (0-10)

SECONDARY OUTCOMES:
Distension after colonoscopy | Change from abdominal distension after the colonoscopy at 20 minutes after.
  Assesment of abdominal distension after colonoscopy by using numerical comparison scale (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.